CLINICAL TRIAL: NCT06415448
Title: Donidalorsen Expanded Access Program for Patients With Hereditary Angioedema (HAE)
Brief Title: Donidalorsen Expanded Access Program for Patients With Hereditary Angioedema
Status: Available | Type: Expanded Access
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISIS 721744-E01
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Angioedema
Keywords: HAE; IONIS PKK-LRx; Donidalorsen; ISIS 721744
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — donidalorsen; IONIS-PKK-LRx

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Donidalorsen — Donidalorsen administered once monthly or every other month by subcutaneous (SC) injections in the abdomen, thigh, or upper arm.
  Other Names: IONIS PKK-LRx; ISIS 721744

SUMMARY:
The purpose of the Expanded Access Program is to provide pre-approval access of donidalorsen to eligible patients with Hereditary Angioedema (HAE) who complete the ISIS 721744-CS3 clinical trial.

DETAILED DESCRIPTION:
The Expanded Access Program (EAP) is intended to provide pre-approval access to donidalorsen for eligible patients with HAE who complete the ISIS 721744-CS3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the ISIS 721744-CS3 (Open-Label Extension [OLE] Study) who have completed 205 weeks of treatment.
* Female patients of childbearing potential, and male patients with partners of childbearing potential must be willing to use acceptable contraception, or refrain from sexual activity.

Exclusion Criteria:

* Any patient who is pregnant or plans to become pregnant.
* Any patient who was withdrawn from the ISIS 721744-CS3 OLE study due to a serious adverse event (SAE) related to donidalorsen therapy or who voluntarily withdrew prior to 205 weeks of treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Related Info — https://www.ionispharma.com/patients/expanded-access-policy/